CLINICAL TRIAL: NCT03374514
Title: Clinical Trial on Cochlear Electrical Impedance and the Effect of Topical Dexamethasone on Cochlear Implant Surgery: The Cochlea as a Capacitor
Brief Title: Cochlear Electrical Impedance and the Effect of Topical Dexamethasone on Cochlear Implant Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, FEDERICO ALBERTO DI LELLA, IP, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3233
Record Dates: First submitted 2017-11-23; First posted 2017-12-15 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Sensorineural Hearing Loss; Cochlear Implant
Keywords: corticosteroids; Electric impedance
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: randomized, controlled and double-blind experimental study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DEX (Experimental): Topical dexamethasone will be placed at a concentration of 20mg / ml in a single dose in the tympanic cavity of the middle ear through posterior tympanotomy in the cochlear implant surgery, paying special attention to the round window membrane completely submerged in the liquid, to the insertion of the electrode assembly
  Interventions: Drug: Dexamethasone
- SF (Placebo Comparator): Sterile isotonic saline solution will be placed in a single dose in the tympanic cavity of the middle ear through posterior tympanotomy during cochlear implant surgery, paying special attention to the fact that the round window membrane is completely submerged in the liquid, prior to insertion of the electrode array
  Interventions: Drug: Sterile isotonic saline solution

INTERVENTIONS:
Drug: Dexamethasone — instilation of the solution in the middle ear
  Arms: DEX
Drug: Sterile isotonic saline solution — Sterile isotonic saline solution
  Arms: SF

SUMMARY:
Hearing is the ability to perceive sounds through the ear. If the transmission of sound is defective, the person suffers some degree of hearing loss. Cochlear Implants (CI) provide partial hearing by stimulating auditory nerve cells.

The evaluation of the functionality of the CI is facilitated by several analysis tools, such as the clinical calibration software. This offers the possibility of measuring electrical impedances in the cochlea. The electrical impedance is the opposition to the current flow between two electrodes. It is composed of two main elements: resistance and reactance. The impedances in a cochlear implant are not stable over time. The value is minimal immediately after surgery, and increases progressively in the first 2 to 3 weeks after the procedure due to the immune response of the organism against a foreign body and the trauma of the array insertion. Several authors have suggested the use of topical or intravenous corticosteroids to decrease intracochlear fibrosis. The use of Dexamethasone could have a protective effect by reducing the initial inflammatory response, apoptosis, and delayed fibrosis, which could impact the impedance.

There is limited evidence on the effect of intra-surgical topical corticosteroids on the impedance of the cochlear implant.

The aim of this clinical trial is to evaluate the impact of topical dexamethasone on the electrical impedance of the cochlear implant, with special attention to the analysis of the capacitive component. It will be carried out through an experimental, prospective, randomized and double-blind study.

Objective To determine whether the use of topical dexamethasone in a single dose applied in the tympanic cavity (middle ear) during cochlear implant surgery modifies the capacitive component of the electrical impedance of the electrodes in the cochlea before the activation of the cochlear implant.

Material and methods A phase 3 clinical trial will be conducted. The design is a parallel, randomized, controlled and double-blind experimental study.

Expected impact The use of local dexamethasone during cochlear implant surgery would decrease the inflammatory response, improving postoperative impedances.

DETAILED DESCRIPTION:
Hypothesis The use of topical dexamethasone in a single dose applied to the tympanic cavity during cochlear implant surgery modifies the capacitive component of the electrical impedance of the electrodes in the cochlea during the first days of the postoperative period.

goals Primary objective To assess whether the use of topical dexamethasone in a single dose applied to the tympanic cavity (middle ear) during cochlear implant surgery, prior to the insertion of the electrode array in the cochlea modifies the capacitive component of the electrical impedance of the cochlear implant. electrodes in the cochlea before activation of the cochlear implant.

Secondary objectives To assess the safety and efficacy of the use of topical dexamethasone in a single dose in the middle ear cavity during cochlear implant surgery.

To estimate the capacitive component of the electrical impedance of the electrodes in the cochlea on a daily basis, from the day of surgery until the day of switching on, in two groups of patients: experimental and placebo.

Materials and methods Design Phase 3 clinical trial design is an experimental parallel, randomized, controlled, double blind assess the effect of the use of topical corticosteroids on the electrical impedance of the electrodes in the cochlea after surgery will be performed of cochlear implant surgery.

All patients diagnosed with severe to profound sensorineural hearing loss unilateral or bilateral that its pathogenesis and pathophysiology are considered candidates for cochlear implantation, will be evaluated as routine in our service, imaging, audiological and psychological studies. Accomplished and accepted the nomination for the placement of one or two cochlear implants will be offered the opportunity to participate in the protocol.

Patients will be selected and those who accept the invitation to participate, the study will be randomly divided into two groups, an experimental group and a placebo group. Randomization was performed in balanced way with a 1: 1 ratio between the branches. The randomisation list will be in blocks of variable size between 2 and 6.

We will proceed as usual to the cochlear implant surgery, using the same anesthetic technique, surgical approach and surgical procedure in any cochlear implant surgery. Technique worldwide known and accepted as "minimally traumatic cochlear implant surgery" (see section definitions below) is used.

The two study groups are:

Group Dexamethasone(DEX):topical administration of dexamethasone (20 mg / ml) in the eardrum of the middle ear through the back tympanostomy, single dose during cochlear implant surgery, prior to inserting the array of electrodes.

Group Placebo / Solution Physiological(SF):topical administration of isotonic sterile physiological solution in the eardrum of the middle ear through the back tympanostomy,single dose during cochlear implant surgery, prior to insertion of the array of electrodes .

After inserting the electrode array into the cochlea, proceed as usual measurements of the electrical responses Intraoperative routine and supplemented with the closure and local healing.

From the date of the surgical procedure and until the final activation of the implant (usually 30 days), you will be asked the patient or family, you make two daily measurements of the impedances of the electrodes, for which he was trained during the hospitalization the day of surgery, the use of a simple software to be distributed for this purpose (CIDC -see later-). The software installed on the computer from the patient can communicate through the common communication interface Cochlear POD (used in clinical practice for starting and calibration of the cochlear implant by the audiologist) and a speech processor Cochlear Freedom (delivered consignment for the study) the implanted device (receiver-stimulator) in patient surgery.

With this software data electrode impedance will be obtained twice a day, in different configurations stimulation and measurement, and will be sent automatically via Internet to a remote server managed by the authors of this protocol.

Postoperative controls on floor and then not differ outpatient than usual for these procedures.

Blind:blind will be maintained for this study the researcher, the patient, evaluation of results and analysts. The only not blind will be who prepares the medication from pharmacy. Electrical impedance measurements are automatic and blind although objective measurements are discussed.

Blind opening procedure:opening blind held immediately in the event of occurrence of an intra or postoperative complication (eg intraoperative hemodynamic alteration, uncontrollable bleeding, infection, fever, allergic reaction, wound dehiscence). Similarly, the blind will be opened for the group of principal investigators, always after completing the stage of implementation of the protocol in patients in question, and each not less than 2 months and the sole purpose of making a partial analysis the results that may involve changing the acquisition parameters of samples for a better interpretation of the results and to fulfill the main objective stipulated.

Place work Patients will be evaluated at the Department of Otolaryngology, Hospital Italiano de Buenos Aires as usual in this type of evaluation. Surgery is carried out in the central operating room of the hospital by any of the three surgeons otologists privileges for these procedures and not differ from the usual surgical technique for cochlear implantation. THe postsurgical controls will be performed in the same service by the same professionals. Measurements of proposals impedances are performed for the oun paciente or his parents, using the same technique and the same equipment used by Audiologists in visits calibration cochlear implants, with help of software designed by researchers specifically for this purpose. The data will be transferred remotely through a security protocol to a fund administered by the principal investigators (cloud) server. Further analysis of the data, evaluation of the results and conclusions of the work will be performed by the principal investigators of this protocol in the field of Hospital Italiano de Buenos Aires.

Population All cochlear implant candidates who meet all inclusion criteria and no exclusion criteria patients and to accept participation in the protocol will be recruited.

Note: If a patient is candidate for bilateral cochlear implant or for the duration of the study is candidate for reimplantation each ear will be considered separately. In this case each ear will be randomized separately following the same procedure.

Definitions Gusher:outpour of perilinfa before the surgical opening of the inner ear.

Minimally traumatic cochlear implant surgery:surgical procedure for placing an electronic implantable device to partially restore hearing function in patients diagnosed with severe sensorineural hearing loss to profound unilateral or bilateral that do not respond to other forms of hearing rehabilitation and meet medical, audiological, radiological and psychological criteria for cochlear implantation.

Minimally traumatic surgical technique consisting placing the receiver-stimulator implant beneath the skin on the temporo-parietal region and an array of electrodes that must be positioned in the scala tympani of the cochlea, not generating any damage to structures level the outer and middle ear (tympanic membrane, middle ear bones) as well as minimum damage to the delicate microstructures inner ear, avoiding maneuvers abrupt opening of the inner ear, suction labyrinthine liquid inlet bone powder or blood the cochlea, and allowing the introduction of the electrode array into the cochlea very slowly, in the direction with better orientation and parallel basal turn the scala tympani.

To do this, the procedure is performed under general anesthesia through a small incision, extending from the tip of the mastoid to temporo-parietal region. It said incision includes the skin, subcutaneous tissue, muscle and periosteum in the same line. A small postero-superior subperiosteal pocket where it will be hosted the receiver-stimulator implant is then generated; for which bone cutter in a small bowl of about 2 cm in diameter. Then a simple mastoidectomy is performed, exposing and preserving the anvil and the approach is completed with a posterior tympanotomy or approach to facial recess under monitoring of the facial nerve and preserving the structure. Ideally it identifies and preserves cord tympani nerve (anterior posterior limit of the tympanostomy). Through the latter the tympanic box is displayed and the round window niche (anatomical repair in relation to the scala tympani of the cochlea) is identified. Careful hemostasis is performed and the mucosa of the margins of the round window DeCola. Usually at this point is necessary and milling at low speed gently and above upper lip of said recess to allow better visualization of the round window membrane (eardrum side). At this point,is necessary for a thorough washing of entire surgical area in order to clear debris or blood bone powder. Then isotonic saline (SF group) or dexamethasone (DEX group) in the tympanic cavity through the posterior tympanotomy, taking special care to the round window membrane is completely submerged in the liquid instill. The implantable device (cochlear implant) is then placed and secured by a suture. At this time it will proceed to the delicate opening of the membranous labyrinth, either through the round window itself, through a small anterior and lower extension thereof or through a cochleostomy (anterior and inferior bone milling margins the round window), performing the endosteal and carefully opening the membranous labyrinth, with special emphasis on not allow entry of bone dust or blood, as well as preventing aspiration of labyrinthine fluid (perilymph). It shall then be slow and progressive introduction of the array of electrodes, with the technique described by the manufacturer as the electrode toused, CI512, CI522 and CI532, progressing the array in the right direction (tangential to the direction of the scala tympani at level of the basal turn of the cochlea) until the entire array of electrodes is positioned within the cochlea. To be completed by sealing the edges of the round window with a small piece of muscle, bone powder level back tympanostomy and finally rearranged the remaining wires in the mastoid cavity, avoiding excessive mobilization, fixing them with a piece of gel foam inside it. The layered closure, periosteum, muscle-fatty cellular and skin absorbable suture is completed. A local flat cure furacinada gauze and a bandage is made. He shall carry out the routine tests and neural response telemetry. End of the surgical procedure.

Intervention Patients admitted with diagnosis of severe sensorineural hearing loss or profound unilateral or bilateral that are evaluated and meet the criteria for candidacy for cochlear implant and comply turn all the inclusion criteria and none of exclusion, will be invited to participate in the study.

Accepted this, a randomized double blind study where the pharmacy is responsible for randomizing treatment among participants proposed subjects. Each of these activities will be properly recorded in writing.

Then they are subjected to usual for placement cochlear implant according the technique of minimally traumatic cochlear implant surgery and used worldwide spread surgery. Reached the operating time in which the round window is displayed (reference anatomical structure of the inner ear and where (or margins) cochlear implant is usually introduced) will proceed as follows, identical in both groups Experimental (DEX) topical dexamethasone (Decadron shock are placed® laboratory Sidus)in concentration of 20mg / ml in single dose in the eardrum of the middle ear through posterior tympanostomy during cochlear implant surgery, taking special care that the membrane round window is completely submerged in the liquid, prior to insertion of the array of electrodes.

Placebo group (SF):

physiologic solution is placed isotonic sterile single dose in the eardrum of the middle ear through posterior tympanostomy during cochlear implant surgery, taking special care that the membrane of the round window is completely submerged in the liquid, prior to insertion of the array of electrodes.

Pharmacy Hospital Italiano de Buenos Aires will be responsible for providing the drug and placebo. It handle it, receiving, contabilizándola, storing and delivering relieving against medical prescription. It will ensure that it is used solely for the purposes of the study. Each of the activities will be recorded in writing. Pharmacy Hospital Italiano de Buenos Aires (HIBA) is the only non blind study participant.

After the surgical procedure, the patient remain hospitalized 24 hours as usual in this type of procedure. Finally cures and weekly inspections shall be made during the first month until activation of the implantable device and continue audiological rehabilitation therapy.

From the day of surgery including, until day programmed for activating the implant, all patients enrolled the study (2 intervening groups) made identically and by themselves or by the help of a relative or guardian, measurements daily (morning and evening) of the impedances of the electrodes of the implant with the CIDC software (available free the day of surgery) and the communication interface POD through a speech processor Cochlear Freedom delivered on consignment during tests for such end.

The result of the measurements of each patient will be sent automatically and as soon as become available internet connection, from the patient's own computer to a remote server (cloud) administered by researchers.

The study ends on the final activation of cochlear implant (approximately 30 days after surgery), at which the implant is permanently connected by the audiologist to your speech processor and the items delivered on consignment for the study will be returned (POD communication interface and speech processor Cochlear Freedom).

Sampling and sample calculation All patients who meet the inclusion criteria and no exclusion to participate in the study and these will be distributed in a randomized into one of two treatment arms will be invited. Monitoring each patient shall be performed within 30 days; it coincides with the usual postoperative controls first week and first postoperative month.

The cochlea with fibrosis exhibit electrical impedance at about 20 KQ compared to a normal cochlea at the day of implant activation (approximately 30 days) 7 KQ with a common standard deviation of 1,481KΩ. To test the null hypothesis that the impedance is equal in patients who were administered steroids and those not were applied, with a power of 80% and an alpha of 5% to test two tailed required 10 patients per group.

With the sample size reached 4980 capacitance values are obtained per patient (20 patients, with 22 electrodes each evaluated in four sequences impedances, with two daily measurements for 30 days). This sample size achieved in 10 patients per group is sufficient for the purpose of describing the behavior of the capacitive impedance component with and without corticosteroid over time.

The sample calculation was performed using STATA 14.0 software and Power and Precision version 4.

Implementation of the clinical

The protocol is conducted in two stages:

Stage 1: Validation "in silico" software to measure impedances. In order to obtain the samples needed to analyze and meet the objectives in this protocol, it is required perform in the patient impedances measurements through the implanted recent device. This is done conventionally in the clinic, by transient connecting a measuring coil which is coupled to implantable device, and through communication interface is integrated to a computer (in the same way that the audiologist makes calibrations sessions on and calibration). By suitable software, measurements can be obtained. However, given the cumbersome and likely poor adhesion to it if you consider that the patient must attend twice a day to treating facility during the first postoperative to make the necessary measurements month, the group of leading researchers this protocol devised and developed their own software that allows a safe, outpatient basis, and the patient's home, taking measurements by himself. In turn, the software in question should allow to measure with the stipulated parameters and the set sequences. The software, called "Cochlear Implant Data Collector (CIDC)" was developed specifically for the realization of this work (and possibly future) and validated by the authors. It is intended to be distributed for free, and installed on the computer from the patient to make measurements. Details thereof, its operation, validation and security are further described in Annex 3.

Step 2: Patient inclusion. Surgery. Impedance measurement Inclusion of patients:Patients who are candidates for cochlear implantation unilateral or bilateral and that meet the selection criteria (see inclusion / exclusion). They explained the protocol and will be asked sign informed consent. It will notify the Hospital Italiano central pharmacy to incorporate the patient randomization and drug preparation / matching placebo for the day of surgery.

Surgical procedure will proceed to the cochlear implant surgery according the conventionally accepted worldwide and known as classic description minimally traumatic cochlear implant surgery (see definitions section). As soon as the access to the tympanic cavity is achieved through the posterior tympanostomy and have identified the round window, proceed according the group randomized to placement or otherwise of the corresponding substance, instilling it directly through the posterior tympanotomy, to completely fill the tympanic cavity, taking special care that the secondary eardrum round window is immersed therein. Then continue with the milling of the bowl to the receiver-stimulator, a cochlear implant is placed in the bed, and slowly and continuously inserting the array of electrodes, either round window round window extended or cochleostomy in ramp will tympanic, according surgeon preference and judgment to meet the primary objective of minimally invasive approach controlling the insertion time in seconds. Finally closing the surgery is completed until completion. It shall then be measuring impedances and neural response as is customary in this procedure.

Measurements using Software "Cochlear Implant Data Collector":out to bring the proposed objective of this study analysis was designed and validated "CIDC" software (see Appendix 3), whereby the patient perform every 12 hs about measurements of the impedances of the electrodes in the sequence routine and established for this purpose in the software.

Sequences stimulation and measurement are as follows:

Sequence1:this sequence involves the monopolar stimulation of each of the 22 intracochlear electrodes as cathode, with the two extracochlear electrodes reference: "Monopolar 1 + 2" (MP1 + 2) Mode (anode). During each stimulation was recorded by measuring the voltage obtained from the same electrode stimulated and reference electrodes in the 14 available time slots by the chipset cic4 implant. Thus 308 samples will be obtained.

Sequence2:Mode "common ground" (CG): this sequence involves stimulation of each of the individual electrodes 22 as cathode, with reference (anode) to the rest of the array of electrodes. During each stimulation was recorded by measuring the voltage obtained between the same electrode and the remaining stimulated intracochlear electrodes in the 14 available time slots by the chipset cic4 implant. Thus 308 samples will be obtained.

Sequence3:Mode "3 points" (3P): intracochlear electrodes will be stimulated sequentially from 1 to 20 inclusive using the following logic: cathode electrode = 'n'; anode electrode = 'n + 2'. Voltage between electrodes nn + 1 is recorded simultaneously at the 14 available time slots by the chipset cic4 implant. Thus 280 samples will be obtained.

Sequence4:Mode "4 points" (4P): intracochlear electrodes stimulate sequentially 1 to 19 inclusive using the following logic: cathode electrode = 'n'; anode electrode = 'n + 3'. The voltage between electrodes n + 1 and n + 2 in the 14 available time slots by the chipset implant cic4 be recorded simultaneously. Thus 266 samples will be obtained.

In each sequence described above is used as stimulation parameters constant the following values:

current level: 80 units of current (corresponding the data sheet chipset cic4 to 74.21 uA) Time between phases: 8 mS Period: 333.4 mS Pulse width : two sequences, 25 and 50 mS

All the sequences described above are made using two different pulse widths predetermined stimulation 25 and 50 mS.

To make these measurements, the company Cochlear LTD or his representative in the country (Tecnosalud SA) provided no cost, a Freedom ™ and an interface POD to connect to computer from the patient, where it install the software processor with a single executable distributed the day of surgery in a pendrive with the appropriate language (Spanish, English, German, Portuguese). All devices will be provided on loan for development work and will be returned to medical team on the day,date on which end data by the patient.

All measured by the software and the context information values (especially the parameters used for each individual measurement and time) are stored in a local database. From the time the application performs periodic attempts to export the data to a database located on a server in the cloud. This database is capable of centralizing measurements unlimited patients. The server is managed and maintained by the principal investigators of this protocol.

Statistical analysis The analysis will be performed by protocol and by intention to treat. The analysis unit be each patient into one of two treatment arms.

Descriptive analysis of quantitative variables with mean and standard deviation or median and interquartile range as observed distribution is expressed. Categorical variables are expressed in proportion to confidence interval for the ratio.

The effect of corticosteroid (dexamethasone) on the variable impedance and capacitance results with generalized equation estimated (GEE) measured. The natural grouping of the individual measurements and the times (panel data) are considered.

Statistical analysis was performed using STATA version 14.0 software. They are considered statistically significant lower probability to 5%.

Clinical management and neglect each patient autonomy be respected to discontinue treatment at any time by communicating to researchers.If the medical staff, researchers or the patient believe that the individual is at risk because the trial, the same will be withdrawn from the study and will explain the reasons why that decision is taken.

Adverse events Adverse events were collected for each control and each time the patient contact the investigator. They are classified according the scale described by Dindo complications and Clavien in 2004 [24,25].Complications are described as deviations from normal postoperative, not including the consequences inherent the procedure itself.

Complications grades are:

Grade 0: no complications Grade I: Any deviation from the normal postoperative course that does not require pharmacological, surgical or endoscopic treatment and does not require radiological interventions. It included in this level using antinauseants, antipyretics, analgesics, diuretics, electrolytes and physiotherapy, as well as drainage of wound infections "bedside".

Grade II: Requires pharmacological treatment with drugs not included in the grade, including transfusions and parenteral nutrition.

Grade III: require surgical, endoscopic or radiological intervention treatment:

IIIa:without general IIIb: anesthesia:general anesthesia Grade IV: life-threatening complication requiring handling unit closed. IVa: Dysfunction of a single body IVb: multiorgan dysfunction Grade V: patient death Damage or complications While complications or damage caused by single topical application of dexamethasone on the round window in single dose during surgery cochlear implant or performing in routine and systematic measurements of the impedances of the electrodes with the proposals and designed in the CIDC software as well as the procedure carried out for measuring them is estimated at zero or extremely rare sequences, the costs of any complications or damages related to procedures or treatments of the study will be funded by the Department of Otolaryngology, Hospital Italiano de Buenos Aires.

Ethical considerations This protocol is drawn and carried in accordance with current national and international standards: Declaration of Helsinki of the World Medical Association, Disposition ANMAT 6770/10 and the Guidelines for Good Clinical Practice ICH E6.

The trial protocol, the patient information and informed consent forms will be submitted to evaluation committee of research projects Hospital Italiano de Buenos Aires (HIBA) (CEPI) for possible approval.

In all cases, the participation of the study is voluntary and certified by the process of informed consent.

The right to opt be respected at all times in the studio without implying in any way any discrimination, differential treatment or abuse without mediate any implication in the treatment of the patient's disease.

Any patient wishing leave the research protocol will be automatically removed from the protocol and not considered for the interpretation of results.

Diagnostic evaluation, surgical procedure, as well as the type, make and model of implantable device used not differ in any way or manner to what is practiced or used routinely in our institution regularly.

All data collected will be treated confidentially and anonymously. Only authorized personnel can access records of study according to the current legal regulation: National Personal Information Protection Law No. 25,326 (Law of Habeas Data).

All patients will be informed of the study objectives; possible adverse events; the procedures; the potential risks they face and; the treatment allocation mechanism. Moreover,is the researcher's responsibility explain to patients their roles in the trial. You will be informed about the strict confidentiality of your personal data, but your medical records may be reviewed for trial purposes by authorized other than your treating physician individuals.

The test results will be stored in accordance with the law of local data protection / ICH GCP - Guidelines and will be treated with utmost confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates to receive a uni or bilateral cochlear implant with diagnosis of severe neurosensory hearing loss.
* Ages between 12 months and 85 years.
* Evaluation of internal ear anatomy performed by tomography and resonance magnetic, where normal cochlea and internal auditory canals are evidenced normal.
* Patients in which any implant of the Cochlear company is used: CI512, CI522 or CI532 with chipset CIC4 or higher.
* Complete insertion of electrodes through round window, round window enlarged or cochleostomy, via posterior tympanotomy using the technique universally known as "minimally traumatic surgery"

Exclusion Criteria:

* Refusal to participate in the protocol or to informed consent
* Intra-surgical gusher (see below, section "definitions").
* Contraindication to receive dexamethasone
* Medical, imaging, psychological or social contraindications to receive a cochlear implant
* Surgical or anesthetic contraindications for cochlear implant surgery.

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
impedance | 30 days
  absolute value
impedance- C | 30 days
  absolute value of the capacitive component
impedance- R | 30 days
  absolute value of the resistive component

CONTACTS AND LOCATIONS:
Locations (1):
- HIBA, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes